CLINICAL TRIAL: NCT06074783
Title: A Patient Sponsored Ongoing Open-label Single-arm, Safety and Efficacy, Phase I/IIb Study of Cellcolabs´ Human Allogeneic Bone-marrow Derived Mesenchymal Stromal Cell Product (StromaForte) in Patients With Musculoskeletal Injuries and/or Degeneration
Brief Title: A Study of Human Allogeneic Bone-marrow Derived Mesenchymal Stromal Cell Product (StromaForte) in Patients With Musculoskeletal Injuries and/or Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellcolabs Clinical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-002-BHS
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Injury
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC Intervention Group (Experimental): Participants will be enrolled into one of four subgroups listed below Firm connective tissue injury (Cartilage, bone, disc, and meniscus) Firm connective tissue degeneration (Cartilage, bone, disc, and meniscus) Soft connective tissue injury (Ligament, tendons, and muscles) Soft connective tissue degeneration (Ligament, tendons, and muscles)
  Treatment: Eligible patients will receive 50 x 106 allogeneic bone marrow (BM)-derived MSC formulated in 4 ml infusion solution of sodium chloride supplemented with human serum albumin to be given locally under ultrasound guidance along with or without 100 x 106 allogeneic BM-derived MSCs formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion in approximately 30 min. Systemic treatment alone is used when local injection at site of injury is not feasible. Additional dose can be administered. Minimum interval between two local doses is 2 months and systemic doses is 3 months.
  Interventions: Biological: Human Allogeneic Bone-Marrow (BM) -Derived Mesenchymal Stromal Cells (MSCs) Product (StromaForte)

INTERVENTIONS:
Biological: Human Allogeneic Bone-Marrow (BM) -Derived Mesenchymal Stromal Cells (MSCs) Product (StromaForte) — 50 x 106 allogeneic BM-derived MSCs formulated in 4 ml infusion solution of sodium chloride supplemented with human serum albumin to be given locally under state of the art way of application that is ultrasound guidance which will ensure precise delivery of the BM derived MSCs at the site of injury or degeneration along with or without 100 x 106 allogeneic BM-derived MSCs formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion in approximately 30 min. Systemic treatment alone is used when local injection at site of injury or degeneration is not feasible.

SUMMARY:
The goal of this ongoing open-label, single-arm, phase I/IIa study in patients is designed to assess the safety of human allogeneic BM-derived MSCs product StromaForte for musculoskeletal injury or/and degeneration. Any male or female with any musculoskeletal injury and/or degeneration above 18 years will be enrolledThe main questions it aims to answer are:

To assess the safety after 28±10, 84±10, 168±10 and 349±10 days of injection by reporting the number of adverse events or severe adverse event assessed by Common Terminology Criteria

Change from baseline in subjective pain assessment in each injured and/or degenerated area (if multiple injury is reported, each area to be followed up separately)

Eligible patients will receive 50 x 106 allogeneic bone marrow (BM)-derived MSC formulated in 4 ml infusion solution of sodium chloride supplemented with human serum albumin to be given locally under ultrasound guidance along with or without 100 x 106 allogeneic BM-derived MSCs formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion in approximately 30 min. Systemic treatment alone is used when local injection at site of injury is not feasible. Additional dose can be administered.

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSDs) and injuries represent a significant global health concern, constituting the primary cause of disability on a global scale. With a high prevalence spanning various stages of life, from childhood to old age, MSDs exert a substantial burden on individuals and society alike. This burden is particularly amplified in the context of an aging population and the prevalence of multi-morbidity. Chronic illnesses and health conditions not only lead to reduced quality of life but also contribute to a substantial financial burden on societies due to increased healthcare costs and lost productivity. In this context, the inability to work and early retirement are often driven by these health issues, forming a critical dimension of the disease burden.

Regular physical exercise is a crucial factor in promoting longevity and overall well-being. Unfortunately, MSDs can significantly impede individuals' ability to engage in exercise and pursue the hobbies and activities that bring them happiness. These disorders often limit mobility, cause pain, and hinder their capacity to lead an active lifestyle.

Addressing and mitigating these MSDs becomes pivotal in restoring individuals' functional capabilities and quality of life. By effectively managing these conditions, we can empower patients to maintain regular exercise routines that contribute to their physical health, mental well-being, and happiness. Encouraging patients to stay active and engaged not only enhances their own lives but also contributes to a healthier and more vibrant society. Ultimately, the ability to exercise and partake in fulfilling activities stands as a cornerstone for longevity, fostering a balanced and fulfilling life journey.

The spectrum of MSDs encompasses a diverse range of conditions, impacting vital musculoskeletal structures such as bones, joints, muscles, tendons, and ligaments [3]. These disorders can originate from a myriad of factors, including traumatic incidents, degenerative processes, autoimmune responses, and genetic predispositions. The consequence is often chronic pain, compromised mobility, diminished physical function, and a diminished quality of life. Among the array of MSDs, the pervasive influence of osteoarthritis is particularly noteworthy, contributing significantly to the global burden of disease.

Addressing musculoskeletal injuries and degeneration presents an urgent imperative due to the widespread prevalence and devastating impact of these conditions. An emerging avenue of exploration lies in the utilization of mesenchymal stem cells (MSCs), which hold immense potential for revolutionizing regenerative medicine. MSCs, found within diverse tissues including bone marrow and adipose tissue, possess the remarkable ability to differentiate into various cell lineages such as osteocytes, chondrocytes, and myocytes. This intrinsic versatility positions them as key players in tissue regeneration and repair.

The rationale for delving into MSC-based therapies rests upon their extraordinary regenerative potential. When applied to the site of injury or degeneration, MSCs can contribute to the reconstitution of damaged tissues, promoting structural and functional recovery. Moreover, MSCs wield immunomodulatory properties, a crucial attribute given the intricate role of the immune response in MSD progression. By modulating immune cell activity, MSCs can foster an anti-inflammatory environment, counteracting the detrimental effects of chronic inflammation observed in numerous MSDs.

In the larger context, the exploration of mesenchymal stem cells as a therapeutic avenue for musculoskeletal injuries and/or degeneration signifies a pioneering leap within the realm of regenerative medicine. The aspiration to alleviate pain, restore mobility, and enhance functionality holds the promise of ameliorating the extensive repercussions endured by individuals grappling with musculoskeletal disorders. MSCs therapy holds the potential to not only alleviate symptoms and improve the quality of life for individuals with musculoskeletal conditions but also to reduce the economic strain caused by decreased workability and early retirement. By promoting tissue repair, reducing inflammation, and enhancing overall musculoskeletal health, MSCs treatment can contribute to extending a person's productive years and lessening the burden on both individuals and society.

Learning more about stem cell applications for a diverse set of musculoskeletal disorders will allow for more specific studies to be designed and more niched groups of study participants to be targeted. A particularly interesting field of indications and study participants resides in the realm of elite sports. Elite athletes, sports teams, organizations, and federations invest huge resources to push the quality in sports to unprecedented levels. In that quest, sports injuries pose a devastating blocker for the athletes and the organizations as it can hamper an individual's career and the success of a team. With this study, one of our aspirations for the future is to partner up with relevant sports associations, teams, and institutions and leverage sought insights to design a study aimed at offering elite athletes the highest quality treatments to help them stay healthy, and in the unlucky event of an injury, return to their sport in the shortest time possible.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and comply with all procedures required by the protocol.
2. Aged ≥ 18 years at the time of signing the informed consent form and has any diagnosed musculoskeletal injury and/or degenerative conditions.

Exclusion Criteria:

1. Unwilling or unable to perform any of the assessments required by the protocol.
2. Have an injury that is expected to selfheal within 14 days without remaining sequel.
3. Have an injury for which there is solid scientific evidence that the study compound will have no effect.
4. Have traumatic head injury or skull, teeth or jaw injury as diagnosis for inclusion in trial.
5. Have an injury that require an orthopaedic surgery that has not been addressed by local/home surgeon.
6. Have end stage liver or renal disease.
7. Have a clinical history of malignancy within 2.5 years (i.e., patients with prior malignancy must be cancer free for 2.5 years) except curatively treated basal cell carcinoma, melanoma in situ, or cervical carcinoma.
8. Have any condition that limits lifespan to < 1 year according to the Principal Investigator's discretion.
9. Hepatitis B virus positive
10. Viraemic Hepatitis C virus, HIV-1/2 or syphilis positive
11. Have unstable angina pectoris, uncontrolled or severe peripheral artery disease within the previous 2 months.
12. Have congestive heart failure defined by New York Heart Association (NYHA) Class IV, or an ejection fraction of <25%.
13. Uncontrolled hypertension (resting systolic blood pressure >220 mm Hg or diastolic blood pressure of > 150 mm Hg at screening) .
14. Have coronary artery bypass surgery, angioplasty, peripheral vascular disease revascularization, or a myocardial infarction within the previous month.
15. Have acute exacerbation of chronic obstructive lung disease stage III or IV (Gold classification), Have cognitive or language barriers that prohibit obtaining informed consent or any study elements.
16. Severe acute infection at time of screening and treatment with study drug
17. Pregnant or Breastfeeding
18. Currently participating (or participated within the previous 30 days of consent) in an investigational therapeutic or device trial.
19. Have a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the patient's participation for the full duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-10-19 (Estimated); Study Completion 2028-10-19 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of human allogenic BM derived MSCs in musculoskeletal injuries and/or degeneration for all patients either face to face or remotely. | From baseline to 1 year
  To assess the safety after 28±10, 84±10, 168±10 and 349±10 days of injection by reporting the number of adverse events or severe adverse event assessed by Common Terminology Criteria For Adverse Events (CTCAE) which is the Incidence of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities determined per the Investigator's judgment for all patients either face to face or remotely.

SECONDARY OUTCOMES:
To evaluate the effect of MSC administration in reported resting pain and pain in movement/loading/weight bearing in each injured and/or degenerated area | From baseline to 1 year
  To evaluate the effect of MSC administration in reported resting pain and pain in movement/loading/weight bearing in each injured and/or degenerated area (if multiple injuries is reported, each area to be followed up separately) from baseline to 28±10, 84±10, 168±10 and 349±10 days for all patients either face to face or remotely.
Change in Health-related quality of life according to Short-Form 36 | From baseline to 1 year
  Change in Health-related quality of life according to Short-Form 36 at 28±10, 84±10, 168±10 and 349±10 days post-injection for all patients either face to face or remotely. SF-36 scores range from 0 (worst) to 100 (best) (5).
Change in Health-related quality of life according to Patient Global Impression of Change | From baseline to 1 year
  Change in Health-related quality of life according to Patient Global Impression of Change at 28±10, 84±10, 168±10 and 349±10 days post-injection for all patients either face to face or remotely. The PGIC scale goes from 1 - 7 with 1 being the best positive outcome and 7 the most negative outcome.
Change in pain assessment | From baseline to 1 year
  Change from baseline in subjective pain assessment. Both resting pain and pain in movement/loading/weight bearing will be assessed according to the VRS questionnaire in pre-existing degenerative disorders, distinct from the condition being treated from the baseline to 28±10, 84±10, 168±10 and 349±10 days for all patients either face to face or remotely. The VRS score is measured 0 - 3 with 0 being no pain and 3 being the maximal pain.
Changes in pain between different treatment subgroups | From baseline to 1 year
  Difference in changes from baseline in pain between subgroups of subjects receiving distinct number of doses at different time intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Live Well, Nassau, The Bahamas, The Bahamas

IPD SHARING:
Plan to Share IPD: Undecided